CLINICAL TRIAL: NCT00943800
Title: Combined Haploidentical-Cord Blood Transplantation for Adults and Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14736B
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Results first posted 2020-10-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Leukemia; Myelodysplastic Syndrome; Multiple Myeloma; Lymphoma
Keywords: Appropriate candidate for transplantation; An HLA-identical related or unrelated donor cannot be identified within an appropriate time frame.
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Multiple Myeloma; Lymphoma | interventions — thymoglobulin; Stem Cell Transplantation; fludarabine; Thiotepa; Antilymphocyte Serum; Whole-Body Irradiation; Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Good Risks patients (Experimental): For patients transplanted in remission.
  Interventions: Drug: Fludarabine-Melphalan & Rabbit antithymocyte globulin (r-ATG); Procedure: Stem Cell Transplant; Procedure: Stem Cells Collections
- High Risk Patients eligible for radiation (Experimental)
  Interventions: Procedure: Stem Cell Transplant; Procedure: Stem Cells Collections; Drug: Fludarabine, Thiotepa, Antithymocyte globulin (ATG), and Total Body Irradiation (TBI)
- High Risk Patients not eligible for radiation (Experimental)
  Interventions: Procedure: Stem Cell Transplant; Procedure: Stem Cells Collections; Drug: Fludarabine, Busulfan, and ATG

INTERVENTIONS:
Drug: Fludarabine-Melphalan & Rabbit antithymocyte globulin (r-ATG) — Fludarabine is given through the vein daily for 5 days. Melphalan is given through the vein daily for 2 days. ATG is given every day in the vein for four days.
  Arms: Good Risks patients
Procedure: Stem Cell Transplant — Infusion of haploidentical donor, umbilical cord blood
Procedure: Stem Cells Collections — Haploidentical cells will be T-cell depleted using the Miltenyi Clinimax device.
Drug: Fludarabine, Thiotepa, Antithymocyte globulin (ATG), and Total Body Irradiation (TBI) — Fludarabine is given through the vein daily for 5 days. Thiotepa is given through the vein daily for 2 days. ATG is given through the vein every other day for 4 days. TBI is given twice a day for 3 days.
  Arms: High Risk Patients eligible for radiation
Drug: Fludarabine, Busulfan, and ATG — Fludarabine is given through the vein daily for 5 days. Busulfan is given through the vein daily for 4 days. ATG is given through the vein every other day for 4 days.
  Arms: High Risk Patients not eligible for radiation

SUMMARY:
The primary objective is to assess the rate of engraftment with combined haploidentical-cord blood transplantation. The secondary objective is to evaluate the incidence and severity of acute and chronic graft-versus-host disease (GVHD).

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for this study if they have any one of the diseases that are known to be cured after allogeneic stem cell transplantation.

1. Relapsed or refractory acute leukemia (myeloid or lymphoid)
2. Acute leukemia in first remission at high-risk for recurrence
3. Chronic myelogenous leukemia in accelerated phase or blast-crisis
4. Chronic myelogenous leukemia in chronic phase
5. Recurrent or refractory malignant lymphoma or Hodgkin lymphoma
6. Chronic lymphocytic leukemia, relapsed or with poor prognostic features
7. Multiple myeloma
8. Myelodysplastic syndrome
9. Chronic myeloproliferative disease
10. Hemoglobinopathies
11. Aplastic anemia

Exclusion Criteria:

1. Zubrod performance status > 2
2. Life expectancy is severely limited by concomitant illness
3. Patients with severely decreased LVEF or impaired pulmonary function tests(PFT's)
4. Estimated Creatinine Clearance <50 ml/min
5. Serum bilirubin> 2.0 mg/dl or SGPT >3 x upper limit of normal
6. Evidence of chronic active hepatitis or cirrhosis
7. HIV-positive
8. Patient is pregnant
9. Patient or guardian not able to sign informed consent

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2006-10-09 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hongtao Liu, M.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Result] Liu H, Rich ES, Godley L, Odenike O, Joseph L, Marino S, Kline J, Nguyen V, Cunningham J, Larson RA, del Cerro P, Schroeder L, Pape L, Stock W, Wickrema A, Artz AS, van Besien K. Reduced-intensity conditioning with combined haploidentical and cord blood transplantation results in rapid engraftment, low GVHD, and durable remissions. Blood. 2011 Dec 8;118(24):6438-45. doi: 10.1182/blood-2011-08-372508. Epub 2011 Oct 5. PMID 21976674
- [Derived] van Besien K, Hari P, Zhang MJ, Liu HT, Stock W, Godley L, Odenike O, Larson R, Bishop M, Wickrema A, Gergis U, Mayer S, Shore T, Tsai S, Rhodes J, Cushing MM, Korman S, Artz A. Reduced intensity haplo plus single cord transplant compared to double cord transplant: improved engraftment and graft-versus-host disease-free, relapse-free survival. Haematologica. 2016 May;101(5):634-43. doi: 10.3324/haematol.2015.138594. Epub 2016 Feb 11. PMID 26869630

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Although the protocol initially had different disease intensities, ultimately, moved to one regimen for all patients.
  Subjects received 30mg/m^2 of Fludarabine from Day-7 until Day-3, 140mg/m^2 of Melphalan on Day-2, and 1.5mg/kg of Rabbit antithymocyte globulin at Day-7,-5,-3 and -1."
Period: Overall Study
Arm/Group | Treatment Group
Started | 87
Completed | 87
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 87
Age, Continuous [Mean (Full Range); unit: years] | 45.5 [10 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 53
  More than one race | 0
  Unknown or Not Reported | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Neutrophil Engraftment
Description: Cumulative incidence of graft failure (neutrophil) by day 28 was reported. Patients who did not have neutrophil engraftment before death was considered as a competing risk. Failure to engraft was defined as lack of evidence of hematopoietic recovery (ANC <500/mm3 and platelet count < 20,000/mm3) by day +35, confirmed by a biopsy revealing a marrow cellularity < 5%. Graft failure was also defined as initial myeloid engraftment by day +35, documented to be of donor origin, followed by a drop in the ANC to < 500/mm3 for more than three days, independent of any myelosuppressive drugs, severe GVHD, CMV, or other infection.
Time Frame: Transplant (Day 0) through Day +28
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment Group
Number analyzed (Participants) | 87
percentage of patients | 85.1 [75.4 to 91.1]

2. Secondary Outcome: Percentage of Participants With Incidence of Acute (Grade II-IV) and Chronic Graft-vs-host Disease(GVHD)
Description: Acute GVHD is defined by the Przepiorka criteria, which stages the degree of organ involvement in the skin, liver, and gastrointestinal (GI) tract, based on severity, with Stage 1+ being least severe and stage 4+ being the most severe. Grading of acute GVHD is as follows: Grade II (skin involvement stages 1+ to 3+, liver 1+, GI tract 1+), Grade III (skin involvement stages 2+ to 3+, liver 1+, GI tract 2+ to 4+), Grade IV (skin involvement stages 4+, Liver 4+).
  Chronic GVHD is assessed by NIH consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant. 2005; 11:945-56., for grading criteria. (See Citation: Filipovich AH et al)
  The incidence of patients with acute GVHD (Grade II-IV) was determined at 180 days. The incidence of Chronic GVHD by 2 years was reported
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment Group
Number analyzed (Participants) | 87
percentage of patients
  Acute GVHD (grade II-IV) | 16.1 [9.3 to 24.6]
  Chronic GVHD | 3.4 [0.9 to 9.0]

3. Secondary Outcome: Overall Survival- Percentage of Participants Who Survived at 2 Years and 5 Years
Description: We reported overall survival at 2 years and 5 years after transplant
Time Frame: up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment Group
Number analyzed (Participants) | 87
percentage of patients
  Two-year overall survival | 43.7 [34.4 to 55.4]
  Five-year overall survival | 32.9 [24.3 to 44.5]

ADVERSE EVENTS:
Time Frame: 100 days
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 18/87
Serious Adverse Events (participants affected / at risk) | 24/87
Other Adverse Events (participants affected / at risk) | 0/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=87)
Abdominal infection (Infections and infestations) | 2
Anemia (Blood and lymphatic system disorders) | 1
Cytokine release syndrome (Immune system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Epstein-barr virus infection (Infections and infestations) | 3
Esophageal infection (Infections and infestations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (Gastrointestinal disorders) | 1
Gait disturbance (General disorders) | 1
Heart failure (Cardiac disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Lung infection (Infections and infestations) | 2
Neutrophil count decreased (Investigations) | 1
Pericardial tamponade (Cardiac disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Sepsis (Infections and infestations) | 11
Skin infection (Infections and infestations) | 1
White blood cell decreased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-12-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT00943800/Prot_SAP_000.pdf